CLINICAL TRIAL: NCT06450873
Title: A Phase 2 Pilot Window of Opportunity Study Turkey Tail Mushrooms (TTM) (Trametes Versicolor) in Post-Menopausal Women With HER2 (-) ER (+) Breast Cancer Planning to Undergo Surgical Therapy
Brief Title: Turkey Tail Mushroom for Treating Post-Menopausal Women With HER2-Negative ER-Positive Breast Cancer Undergoing Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC220305; NCI-2024-03999 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-003846 (Other: Mayo Clinic Institutional Review Board); MC220305 (Other: Mayo Clinic)
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Estrogen Receptor-Positive Breast Carcinoma; HER2-Negative Breast Carcinoma
MeSH Terms: interventions — VPS Coriolus versicolor extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (TTM) (Experimental): Patients receive TTM PO BID starting at the time of study registration and continuing up to the day prior to SOC surgery (up to 3-6 weeks) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Coriolus Versicolor Extract; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Coriolus Versicolor Extract — Dietary Supplement Given PO
  Other Names: Turkey Tail Mushroom Extract; Yunzhi Extract
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial tests how well turkey tail mushroom (TTM) works in treating post-menopausal women with HER2-negative, estrogen receptor (ER)-positive breast cancer undergoing surgery. TTM is a common mushroom. In traditional Chinese medicine, it is used for enhancing function and removing toxins, as well as for cancer, hepatitis, and infections. There is previous evidence of significant tumor shrinkage occurring in the 2-month window between diagnosis and surgery in women who have taken TTM. Giving TTM may be effective in treating post-menopausal women with HER2-negative, ER-positive breast cancer undergoing surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine changes in proliferation (Ki-67) in ER+HER2- breast cancers that receive turkey tail administration.

SECONDARY OBJECTIVES:

I. To assess associated adverse effects of coriolus versicolor extract (TTM). II. To determine if quality of life (QOL), mood and energy levels change while taking TTM.

OUTLINE:

Patients receive TTM orally (PO) twice daily (BID) starting at the time of study registration and continuing up to the day prior to standard of care (SOC) surgery (up to 20-42 days) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up 7-30 days after last dose.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years of age
* Histological confirmation of ER+, HER2- breast cancer, newly diagnosed and tissue available for central confirmation of Ki-67 measurement. Ki-67 will be repeated for patients who have had this done externally.
* Scheduled for definitive breast surgery
* Detectable disease as defined by mammography, breast ultrasound of greater than 5mm in size.

  * NOTE: Tumor lesions in a previously irradiated area are not considered measurable disease; Disease that is measurable by physical examination only is not eligible
* Post menopausal as defined by:

  * Self-reported last menstrual period greater than 12 months, or
  * Bilateral oophorectomy, or
  * Follicle stimulating hormone (FSH) >20 mIU/mL, and estradiol level ≤ 20 pg/mL
* Not taking aromatase inhibitor or a selective estrogen receptor modifier
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2 obtained ≤ 90 days prior to registration
* Platelet count ≥ 100,000/mm^3 (obtained ≤ 90 days prior to registration)
* Absolute neutrophil count (ANC) ≥ 1,000/mm^3 (obtained ≤ 90 days prior to registration)
* Hemoglobin ≥ 11 g/dL (obtained ≤ 90 days prior to registration)
* Serum transaminase [alanine aminotransferase (ALT) or aspartate aminotransferase (AST)] ≤ 1.2 x upper limit of normal (ULN) (obtained ≤ 90 days prior to registration)
* Alkaline phosphatase ≤ 1.2 x ULN (obtained ≤ 90 days prior to registration)
* Serum creatinine ≤ 1.2 x ULN (obtained ≤ 90 days prior to registration)
* Provide written informed consent
* Ability to complete the Symptom Experience Diary by themselves or with assistance

Exclusion Criteria:

* Current use of any medicinal mushrooms
* Patient with locally advanced cancer who will require neoadjuvant therapy or metastatic cancer
* Currently on systemic chemotherapy
* Concurrent endocrine therapy (selective estrogen receptor modifiers or aromatase inhibitors)
* Allergy to mushrooms
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients
* Patients known to be HIV positive and currently receiving antiretroviral therapy.

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy 3 years prior to registration

  * EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix
  * NOTE: If there is a history of prior malignancy, they must not be receiving chemotherapy treatment for their cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Ki-67 | Baseline; at the time of surgery
  Change in Ki-67 from the time of enrollment (pre-treatment) to the time of surgery (post-treatment) will be recorded. Slides from the original biopsy at the time of diagnosis will be used to assess pre-treatment Ki-67. A tissue sample obtained at the time of surgery will be used to assess Ki-67 post-treatment.

SECONDARY OUTCOMES:
Quality of life changes | Up to 10 weeks
  Changes in quality of life will be assessed using the Symptom Experience Diary, which will be completed by study staff during weekly phone calls with participants. The Symptom Experience Diary consists of 2 yes/no questions and 10 questions answered on a scale of 0-10 where 0=none at all and 10=as bad as it can be.
Adverse effects of Turkey Tail Mushrooms (TTM) | Up to 10 weeks
  Adverse effects of TTM will be assessed by the number of patients with grade 2 or higher toxicities.
Patient-reported outcomes | Up to 10 weeks
  Patient reported outcomes will be assessed using the Symptom Experience Diary, which will be completed by study staff during weekly phone calls with participants. The Symptom Experience Diary consists of 2 yes/no questions and 10 questions answered on a scale of 0-10 where 0=none at all and 10=as bad as it can be.

CONTACTS AND LOCATIONS:
Overall Officials: Larry R. Bergstrom, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials